CLINICAL TRIAL: NCT04898088
Title: A Proof of Concept Study for the DNA Repair Driven by the Mesenchymal Stem Cells in Critical COVID-19 Patients
Acronym: REPAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SBÜ Dr. Sadi Konuk Eğitim ve Araştırma Hastanesi (Other)
Collaborators: Istinye University (Other); Liv Hospital (Ulus) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8860/9193
Record Dates: First submitted 2021-05-21; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19; Critical Case; DNA Repair; DAN damage
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Therapy (Experimental)
  Interventions: Biological: Mesenchymal Stem Cells Transplantation
- Conventional Therapy with Add-On MSC therapy (Experimental)
  Interventions: Biological: Mesenchymal Stem Cells Transplantation

INTERVENTIONS:
Biological: Mesenchymal Stem Cells Transplantation — Mesenchymal Stem Cells Transplantation applied as three intravenous infusions with 30 days intervals

SUMMARY:
Our aim in this study is to determine the positive effect of stem cell therapy applied on critically ill patients with coronavirus infection on DNA repair genes.

Patients diagnosed with COVID-19 infection are divided into two equal (n:30) groups. Group-1(n/15): Patients in critically ill condition receiving conventional therapy, Group-2 (n/15): Patients in critically ill condition receiving conventional therapy and systemically transplanted MSCs. The DNA repair pathway will be examined as 11 genes in 5 different parts. Investigated parameters:

1. Base excision repair
2. Nucleotide excision repair
3. Recombinational repair
4. Mismatch repair
5. Direct reversal Investigated parameters: broad biochemical analysis, apoptosis, clinical outcome, and mortality rates.

DETAILED DESCRIPTION:
Our aim in this study is to determine the positive effect of stem cell therapy applied on critically ill patients with coronavirus infection on DNA repair genes.

Patients diagnosed with COVID-19 infection are divided into two equal (n:30) groups. Group-1(n/15): Patients in critically ill condition receiving conventional therapy, Group-2 (n/15): Patients in critically ill condition receiving conventional therapy and systemically transplanted MSCs. The DNA repair pathway will be examined as 11 genes in 5 different parts. Investigated parameters:

1. Base excision repair
2. Nucleotide excision repair
3. Recombinational repair
4. Mismatch repair
5. Direct reversal Investigated parameters: broad biochemical analysis, apoptosis, clinical outcome, and mortality rates.

ELIGIBILITY:
Inclusion Criteria:

1. 40-65 years old male/female.
2. Obtaining informed consent from him or his legal relative.
3. Confirmed COVID-19 related severe ARDS cases.

Exclusion Criteria:

pregnant, malignant tumours, the ones who has confirmed co-infection; history of using long-term immunosuppressive agents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Expression of PARP1 gene as indicator of base excision repair | 6 months
  Expression of PARP1 gene as indicator of base excision repair
Expression of genes ATM, RAD51, RAD52 and WRN as indicator of Recombinational repair | 6 months
  Expression of genes ATM, RAD51, RAD52 and WRN as indicator of Recombinational repair
Expression of genes RAD23B and ERCC1 as indicator of Nucleotide excision repair | 6 months
  Expression of genes RAD23B and ERCC1as indicator of Nucleotide excision repair
Expression of genes MLH1, MSH2 and MSH6as indicator of Mismatch repair | 6 months
  Expression of genes MLH1, MSH2 and MSH6 as indicator of Mismatch repair

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Istinye University, Istanbul
  - SBÜ Dr. Sadi Konuk Eğitim ve Araştırma Hastanesi, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided